CLINICAL TRIAL: NCT01944488
Title: LH Response to GnRH Test in Prepubescent Girls Under 6 Years
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1-10-72-631-12
Record Dates: First submitted 2013-09-06; First posted 2013-09-17 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Precocious Puberty
Keywords: Precocious puberty; GnRH-test
MeSH Terms: conditions — Puberty, Precocious | interventions — Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GnRH intervention (Experimental): All participating subjects are assigned to receive an intravenous GnRH agonist injection.
  Interventions: Drug: GnRH agonist

INTERVENTIONS:
Drug: GnRH agonist — 100 µg/m2 body surface max 100 µg i.v.
  Other Names: LHRH agonist

SUMMARY:
The project aims to establish the normal LH and FSH response to a standardized GnRH dose in healthy girls below 6 years of age, and compares the normal GnRH response to the GnRH response in girls with early puberty development.

The novel data may help to determine whether the girl is in early puberty or not.

Healthy girls under 6 years of age attending routine examinations including an i.v. line for other causes are included in this study. Our examinations also include bone age determination, Tanner stage determination, and anthropometric measures (height and weight). 10 healthy girls in each of the following age groups: 7-12 months, 12-24 months, 24-36 months, 36-48 months, 48-60 months and 60-72 months are included.

DETAILED DESCRIPTION:
Please refer to the brief summary which covers the study aim, methods and outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Endocrinologically healthy girls in the age from 7 months to 6 years
* Obtained oral and written informed consent from participants parents

Exclusion Criteria:

* Anamnestic, clinical or laboratory findings that indicate that the subject is suffering from other diseases (eg poorly controlled asthma) or is in a condition which might affect the subject's ability to complete the study or which is likely to affect the parameters under investigation.
* Current medical treatment apart from prophylactic antibiotics or weak analgesics.
* GFR <50 ml/min/1,73m2 or if absence of previous GFR study: serum creatinine above normal upper age-specific normal range.
* Clinical signs of precocious puberty

Ages: 7 Months to 6 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
LH response | 30 minutes

SECONDARY OUTCOMES:
FSH response | 30 minutes

OTHER OUTCOMES:
Weight | Up till age 6.0 years
Height | Up till age 6.0 years
Tanner-stage (breast and pubic hair) | Up till age 6.0 years
Bone age | Up till age 6.0 years
Hormones (estrogen, inhibin B, SHBG, kisspeptin) | Up till age 6.0 years

CONTACTS AND LOCATIONS:
Overall Officials: Niels H. Birkebæk, MD PhD, Principal Investigator — Børneafdeling A, AUH, Skejby; Esben T. Vestergaard, MD PhD, Principal Investigator — Børneafdeling A, AUH, Skejby; Kurt Kristensen, MD PhD, Principal Investigator — Børneafdeling A, AUH, Skejby; Søren Rittig, MD DMSc, Principal Investigator — Børneafdeling A, AUH, Skejby; Kostas Kamperis, MD PhD, Principal Investigator — Børneafdeling A, AUH, Skejby; Mia E. Sømod, Stud.med, Principal Investigator — Børneafdelig A, AUH, Skejby
Locations (1):
- Børneafdelingen A, AUH, Skejby, Aarhus N, Denmark

REFERENCES:
- [Background] Carel JC, Leger J. Clinical practice. Precocious puberty. N Engl J Med. 2008 May 29;358(22):2366-77. doi: 10.1056/NEJMcp0800459. No abstract available. PMID 18509122
- [Background] Teilmann G, Pedersen CB, Jensen TK, Skakkebaek NE, Juul A. Prevalence and incidence of precocious pubertal development in Denmark: an epidemiologic study based on national registries. Pediatrics. 2005 Dec;116(6):1323-8. doi: 10.1542/peds.2005-0012. PMID 16322154
- [Background] Herman-Giddens ME, Slora EJ, Wasserman RC, Bourdony CJ, Bhapkar MV, Koch GG, Hasemeier CM. Secondary sexual characteristics and menses in young girls seen in office practice: a study from the Pediatric Research in Office Settings network. Pediatrics. 1997 Apr;99(4):505-12. doi: 10.1542/peds.99.4.505. PMID 9093289
- [Background] Houk CP, Kunselman AR, Lee PA. The diagnostic value of a brief GnRH analogue stimulation test in girls with central precocious puberty: a single 30-minute post-stimulation LH sample is adequate. J Pediatr Endocrinol Metab. 2008 Dec;21(12):1113-8. doi: 10.1515/jpem.2008.21.12.1113. PMID 19189683
- [Background] Curfman AL, Reljanovic SM, McNelis KM, Dong TT, Lewis SA, Jackson LW, Cromer BA. Premature thelarche in infants and toddlers: prevalence, natural history and environmental determinants. J Pediatr Adolesc Gynecol. 2011 Dec;24(6):338-41. doi: 10.1016/j.jpag.2011.01.003. PMID 22099730
- [Background] Atay Z, Turan S, Guran T, Furman A, Bereket A. The prevalence and risk factors of premature thelarche and pubarche in 4- to 8-year-old girls. Acta Paediatr. 2012 Feb;101(2):e71-5. doi: 10.1111/j.1651-2227.2011.02444.x. Epub 2011 Sep 23. PMID 21854448
- [Background] de Vries L, Guz-Mark A, Lazar L, Reches A, Phillip M. Premature thelarche: age at presentation affects clinical course but not clinical characteristics or risk to progress to precocious puberty. J Pediatr. 2010 Mar;156(3):466-71. doi: 10.1016/j.jpeds.2009.09.071. Epub 2009 Nov 14. PMID 19914634
- [Background] Resende EA, Lara BH, Reis JD, Ferreira BP, Pereira GA, Borges MF. Assessment of basal and gonadotropin-releasing hormone-stimulated gonadotropins by immunochemiluminometric and immunofluorometric assays in normal children. J Clin Endocrinol Metab. 2007 Apr;92(4):1424-9. doi: 10.1210/jc.2006-1569. Epub 2007 Feb 6. PMID 17284632
- [Background] Brito VN, Batista MC, Borges MF, Latronico AC, Kohek MB, Thirone AC, Jorge BH, Arnhold IJ, Mendonca BB. Diagnostic value of fluorometric assays in the evaluation of precocious puberty. J Clin Endocrinol Metab. 1999 Oct;84(10):3539-44. doi: 10.1210/jcem.84.10.6024. PMID 10522992